CLINICAL TRIAL: NCT05276791
Title: Endoscopic Mucosal Resection Versus Endoscopic subMucosal Dissection fOr Removal of Visible Lesions in Barrett's Esophagus With Early Neoplasia: a Randomized Controlled Trial
Brief Title: EMR Versus ESD for Barrett's Neoplasia
Acronym: REMOVE-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: University Medical Center Groningen (Other); Amsterdam UMC, location VUmc (Other); Erasmus Medical Center (Other); UMC Utrecht (Other); Catharina Ziekenhuis Eindhoven (Other); St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Sanne van Munster, Principal Investigator (Bas Weusten), Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2022-03-01; First posted 2022-03-11 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Barretts Esophagus With Dysplasia; Barrett Adenocarcinoma; Esophageal Cancer
Keywords: Barrett's esophagus; Esophagheal adenocarcinom
MeSH Terms: conditions — Esophageal Neoplasms; Barrett Esophagus

STUDY DESIGN:
Intervention Model Description: Randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic submucosal dissection (Active Comparator)
  Interventions: Other: ESD
- Endoscopic mucosal resection (Active Comparator)
  Interventions: Other: EMR

INTERVENTIONS:
Other: EMR — Endoscopic mucosal resection, according to standard care
  Arms: Endoscopic mucosal resection
Other: ESD — Endoscopic submucosal dissection, according to standard care
  Arms: Endoscopic submucosal dissection

SUMMARY:
Rationale:

The optimal technique for removal of visible dysplastic lesions in Barrett's esophagus remains controversial. Endoscopic mucosal resection (EMR) is safe, effective, easy to apply, and has been the most widely used technique since 2008. Endoscopic submucosal dissection (ESD) is a more controlled dissection method with potential improved efficacy, but at the cost of higher technical complexity.

Objective:

The investigators aim to compare EMR and ESD for removal of visible lesions in Barrett's esophagus.

Study design:

Randomized clinical trial

Study population:

Patients with Barrett's esophagus and a visible lesion with dysplasia and/or early cancer. Suspicion for submucosal invasion is an exclusion criterion.

Intervention:

Patients are randomized to receive either EMR or ESD, with follow-up and no ablation during 12 months after the resection.

Main study endpoint:

Primary endpoint is the proportion of patients with no evidence of residual or local recurrent neoplasia during 12 months follow-up after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients age: ≥ 18 years
* Willingness to undergo both EMR or ESD
* Ability to provide written, informed consent (approved by IRB) and understand the responsibilities of trial participation
* BE with a single visible lesion with absence of signs of submucosal invasion on endoscopy, after evaluation by the adjudication committee.

Exclusion Criteria:

* Patients with visible lesions with suspicion of submucosal invasion bases on assessment of the adjudication committee
* History of esophageal surgery other than fundoplication
* History of esophageal ablation therapy or endoscopic resection
* Multiple visible lesions in the BE segment at baseline
* Uncontrolled coagulopathy with INR >2.0, thrombocytopenia with platelet counts < 50,000
* Subject has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment in-structions, or follow-up guidelines
* Life expectancy <2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint is the proportion of patients with no evidence of residual or local recurrent neoplasia during 12 months follow-up after baseline. | 12 months

SECONDARY OUTCOMES:
Incidence of complications | 12 months
  . Complications will be assessed on patient level (yes/no) and chi-square test will be used to compare the outcomes between the study arms. In the case > 25% of patients have multiple complications, assessment will be performed on complication level (n per patient) using Poisson-regression analysis.
Procedure times | 12 months
  a skewed continuous variable that will be compared using the Mann-Whitney U test.
Proportion of patients with endoscopically radical resection | 12 months
  assessed during the ER endoscopy, a proportion that will be compared using the chi2 test or Fisher's exact if the number of patients in a single category is <5.
The total number of ER endoscopies per patient | 12 months
  This number will be compared using Poison regression analysis.
The proportion of patients that shows neoplastic progression | 12 months
  This will be compared with a chi2 test or Fisher's exact if the number of patients in a single category is <5, and this analyses will be stratified for moment of detection (i.e. at baseline or later during the study duration).
Cost-effectiveness | 12 months
  Cost-effectiveness will be calculated by efficacy of both procedures (absence of residual or recurrent disease) divided by total costs in Euro associated with the procedures
Additional histopathologic evaluation may be performed to evaluate potential differences between the two techniques. | 12 months
  Interobserver agreement between the two techniques will be evaluated with Cohen's kappa, as well as a subjective score on ease of assessment on a NRS score ranging from 0-10.

IPD SHARING:
Plan to Share IPD: No